CLINICAL TRIAL: NCT03298633
Title: Intracytoplasmic Sperm Injection (ICSI) Versus Conventional in Vitro Fertilization (IVF) in Couples With Non-severe Male Infertility: a Randomized Controlled Trial
Brief Title: ICSI Versus Conventional IVF in Couples With Non-severe Male Infertility
Acronym: ICSI/IVF-NSMI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jie Qiao (Other)
Collaborators: International Peace Maternity and Child Health Hospital (Other); Women's Hospital School Of Medicine Zhejiang University (Other); Sixth Affiliated Hospital, Sun Yat-sen University (Other); First Affiliated Hospital of Kunming Medical University (Other); Beijing Haidian Maternal and Child Health Hospital (Other); The First Affiliated Hospital of Anhui Medical University (Other); The Second Hospital of Hebei Medical University (Other); The Third Affiliated Hospital of Guangzhou Medical University (Other); General Hospital of Ningxia Medical University (Other)
Responsible Party: Sponsor-Investigator, Jie Qiao, President, Peking University Third Hospital
Organization: Peking University Third Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ICSI/IVF-NSMI
Record Dates: First submitted 2017-09-22; First posted 2017-10-02 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Male Infertility
Keywords: Male infertility; In vitro fertilization; Intracytoplasmic sperm injection
MeSH Terms: conditions — Infertility, Male | interventions — Sperm Injections, Intracytoplasmic

STUDY DESIGN:
Intervention Model Description: Eligible patients that have provided informed consent will be randomized to either ICSI or conventional IVF. Randomization and allocation of patients to study groups will be performed on the day of oocyte retrieval. Stratified permuted block randomization will be centrally controlled by administrative staffs in the trial center, who are not involved in the treatment procedure. When there is an eligible participant to be enrolled into the study, nurses from the specific site will login the trial system to get allocation of patients according to a computer-generated randomization list in a 1:1 ratio, with a variable block size of 2, 4 or 8 and stratified by center.
Masking Description: The blinding method in out study is open-label in general. However, in order to avoid psychological effect for participants and unexpected drop-off, the trial is designed to inform participants their insemination method on the day of fresh embryo transfer or the day of embryo freezing. Prior to this, randomization will be strictly performed and keep secret to participants and clinicians.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intracytoplasmic Sperm Injection (Active Comparator): On the day of oocyte retrieval, qualified participants will be randomized into either of two groups. Participants in group A will undergone Intracytoplasmic Sperm Injection (ICSI) procedure, other standard assisted reproductive treatments are similar and parallel between two groups.
  Interventions: Other: ICSI
- Conventional IVF (Active Comparator): On the day of oocyte retrieval, qualified participants will be randomized into either of two groups. Participants in this group will undergone Conventional In Vitro Fertilization (IVF) procedure, other standard assisted reproductive treatments are similar and parallel between two groups.
  Interventions: Other: Conventional IVF

INTERVENTIONS:
Other: ICSI — All patients will receive controlled ovarian hyperstimulation (COH) treatment, which is performed by standard routines at each study center. The COH treatment includes either gonadotrophin-releasing hormone agonist (GnRH-a) protocol or gonadotrophin-releasing hormone antagonist (GnRH-ant) protocol.Oocyte retrieval is scheduled for 36 (±2) after hCG injection.The retrieved cumulus oocyte complexes (COC) will be allocated to undergo routine ICSI procedure according to the result of randomization in each study site.
  Arms: Intracytoplasmic Sperm Injection
Other: Conventional IVF — All patients will receive controlled ovarian hyperstimulation (COH) treatment, which is performed by standard routines at each study center. The COH treatment includes either gonadotrophin-releasing hormone agonist (GnRH-a) protocol or gonadotrophin-releasing hormone antagonist (GnRH-ant) protocol.Oocyte retrieval is scheduled for 36 (±2) after hCG injection.The retrieved cumulus oocyte complexes (COC) will be allocated to undergo conventional IVF procedure according to the result of randomization in each study site.
  Arms: Conventional IVF

SUMMARY:
A multicenter, parallel-controlled(1:1 treatment ratio), open-label, randomized clinical trials regarding fertilization and pregnancy outcomes between ICSI and conventional IVF among couples with no-severe male-factor infertility in China.

DETAILED DESCRIPTION:
A multicenter, large-scale, randomized controlled clinical trial will enroll 2,346 couples with non-severe male infertility undergoing their first or second cycle of IVF or ICSI. The study will recruit participants from 6 Reproductive Medical Centers across mainland China.The participation in this study will be approximately 2 years with a total of 7 visits from controlled ovarian hyperstimulation, pregnancy to delivery. On the day of oocyte retrieval, eligible participants will be allocated to two groups at a ratio of 1:1- ICSI protocol, and conventional IVF protocol. All participants will be randomized through stratified block randomization according to the study sites.

ELIGIBILITY:
Inclusion Criteria:

* Infertile couples scheduled for their first or second IVF/ICSI cycle.
* Men with non-severe male infertility: Sperm concentration 5,000,000-15,000,000/ml or sperm with progressive motility (type A+B) 10-32%.
* Women received either gonadotrophin-releasing hormone agonist protocol or gonadotrophin-releasing hormone antagonist protocol as their controlled ovarian hyperstimulation treatment.
* Informed consent obtained.

Exclusion Criteria:

* Couple with contraindication for IVF or ICSI.
* Couples receiving donor sperm or donor eggs.
* Couples undergoing PGD and PGS.
* Sperm concentration with progressive motility used for insemination <100,000/ml on the day of oocyte retrieval.
* Women with 0 oocytes after oocyte retrieval.
* Using frozen semen.
* Poor fertilization in previous cycle (≤ 25%).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2387 (Actual)
Dates: Start 2018-04-04 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Ongoing pregnancy leading to live birth after the first cycle with embryo transfer | After 22 weeks of gestation
  A delivery of one or more living infants (≥22 weeks gestation or birth weight more than 1,000g).

SECONDARY OUTCOMES:
Fertilization | 16-20 hours after oocyte retrieval
  Number of zygotes with 2 PN (per oocyte retrieved and per women randomized).
Total fertilization failure | 72 hours after oocyte retrieval
  No oocyte formed 2 PN in this given cycle.
Available embryo | 72 hours after oocyte retrieval
  Number of embryos ≥4 cells and ≤30% fragmentation on day 3 observation.
Good quality embryo | 72 hours after oocyte retrieval
  Number of embryos with ≥6 cells and ≤30% fragmentation developed from 2PN embryos on day 3 observation.
Implantation | 28 days after embryo transfer
  Number of gestational sacs observed per embryo transferred.
Clinical pregnancy | 7 weeks after embryo transfer
  One or more observed gestational sac or definitive clinical signs of pregnancy under ultrasonography at 7 weeks after embryo transfer (including clinically documented ectopic pregnancy).
Multiple pregnancy | 7 weeks after embryo transfer
  Pregnancy with two or more gestational sacs or positive heart beats at 7 weeks of gestation.
Ongoing pregnancy | 12 weeks after embryo transfer
  Presence of a gestational sac and fetal heartbeat after 12 weeks of gestation.
Moderate/severe ovarian hyperstimulation syndrome (OHSS) | From date of controlled ovarian hyperstimulation until the date of oocyte retrieval, assessed about 14-16 days.
  exaggerated systemic response to ovarian stimulation characterized by a wide spectrum of clinical and laboratory manifestations. It is classified as mild, moderate, or severe according to the degree of abdominal distention, ovarian Enlargement, and respiratory, hemodynamic, and metabolic complications.
Miscarriage | 22 weeks of gestation
  Spontaneous loss of an intra-uterine pregnancy prior to 22 completed weeks of gestational age.
Ectopic pregnancy | 7 weeks of gestation
  Implantation takes place outside the uterine cavity, confirmed by sonography or laparoscopy.
Gestational diabetes mellitus (GDM) | 24-37 weeks of pregnancy
Hypertensive disorders of pregnancy | 28-37 weeks of pregnancy
  Comprising pregnancy induced hypertension (PIH); pre-eclampsia (PET) and eclampsia.
Antepartum haemorrhage | 28-37 weeks of pregnancy
  Including placenta previa, placenta accreta and unexplained.
Preterm birth | 28-37 weeks of pregnancy
  Birth of a fetus delivered after 28 and before 37 completed weeks of gestational age in participants confirmed ongoing pregnancy.
Birth weight | Within 2 weeks after live birth
  Including low birth weight (defined as weight < 2500 gm at birth), very low birth weight (defined as < 1500 gm at birth), high birth weight (defined as >4000 gm at birth) and very high birth weight (defined as >4500 gm at birth).
Large for gestational age | Within 2 weeks after live birth
  Birth weight >90th centile for gestation, based on standardised ethnicity based charts.
Small for gestational age | Within 2 weeks after live birth
  Less than 10th centile for gestational age at delivery based on standardised ethnicity based charts.
Congenital anomaly | Within 2 weeks after live birth
  Any congenital anomaly will be included.
Perinatal mortality | Within 6 weeks after live birth
  Fetal or neonatal death occurring during late pregnancy (at 28 completed weeks of gestational age and later), during childbirth, or up to seven completed days after birth.
Neonatal mortality | Within 6 weeks after live birth
  death of a live born baby within 28 days of birth

CONTACTS AND LOCATIONS:
Overall Officials: Jie Qiao, M.D., Study Director — Peking University Third Hospital
Locations (10):
- China (10):
  - First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Peking University third Hospital, Beijing, Beijing Municipality
  - Haidian Maternal and Child Health Hospital, Beijing, Beijing Municipality
  - The Third Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - The Sixth Affiliated Hospital of Sun Yat-Sen University, Guangzhou, Guangdong
  - The Second Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - General Hospital of Ningxia Medical University, Yinchuan, Ningxia
  - International Peace Maternity and Child Health Hospital of Shanghai Jiao Tong University, Shanghai, Shanghai Municipality
  - First Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - Women's Hospital of Zhejiang University, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang Y, Li R, Yang R, Zheng D, Zeng L, Lian Y, Zhu Y, Zhao J, Liang X, Li W, Liu J, Tang L, Cao Y, Hao G, Wang H, Zhang H, Wang R, Mol BW, Huang H, Qiao J. Intracytoplasmic sperm injection versus conventional in-vitro fertilisation for couples with infertility with non-severe male factor: a multicentre, open-label, randomised controlled trial. Lancet. 2024 Mar 9;403(10430):924-934. doi: 10.1016/S0140-6736(23)02416-9. Epub 2024 Feb 5. PMID 38330980
- [Derived] Zheng D, Zeng L, Yang R, Lian Y, Zhu YM, Liang X, Tang L, Wang H, Cao Y, Hao G, Liu J, Zhao J, Wang R, Mol BW, Li R, Huang HF, Qiao J. Intracytoplasmic sperm injection (ICSI) versus conventional in vitro fertilisation (IVF) in couples with non-severe male infertility (NSMI-ICSI): protocol for a multicentre randomised controlled trial. BMJ Open. 2019 Sep 30;9(9):e030366. doi: 10.1136/bmjopen-2019-030366. PMID 31575574